CLINICAL TRIAL: NCT02721901
Title: Development and Assessment of iEAT for Use by Parents in the Home Setting
Brief Title: Integrated Eating Aversion Treatment Manual-Parent Version
Acronym: iEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William Sharp, PhD, PhD, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00086399
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Feeding and Eating Disorders of Childhood
Keywords: Gastrointestinal Disorders; Nutrition; Behavioral
MeSH Terms: conditions — Feeding and Eating Disorders of Childhood; Gastrointestinal Diseases; Behavior | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iEAT Manual Intervention (Experimental): Caretakers of 10 children will be randomized to participate in the integrated Eating Aversion Treatment (iEAT) intervention. iEAT is a technology-based manual which aims to increase the child's food consumption.
  Interventions: Behavioral: iEAT Manual Intervention
- Control group (Active Comparator): Caretakers of 10 children will be randomized to participate in the control group. Participants assigned to the control group will be able to receive the iEAT treatment after the study ends.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: iEAT Manual Intervention — The iEAT manual guides caretakers in increasing the volume of food consumed by the child. The manual involves a touch screen application that collects and stores data on key behaviors and provides the feeder with direction for structuring treatment meals. Sessions will be 45 minutes long and occur biweekly for 10 sessions over 5 months. Two meals each day will be completed at home as part of the treatment of the feeding problems.
  Arms: iEAT Manual Intervention
Behavioral: Control group — The psychoeducation condition will involve 6 appointments (once monthly for 5 months and 1 session during the post-treatment assessment). Each appointment will include curriculum related to feeding concerns such as the etiology of feeding problems, meal structure, appropriate food selection, mealtime problem behaviors, and generalization of appropriate feeding behaviors. Each session will last approximately 45 minutes.
  Arms: Control group

SUMMARY:
The purpose of this study is to further develop the integrated Eating Aversion Treatment (iEAT) manual, which is designed to address chronic food aversion in children with chronic food refusal. This study will evaluate the feasibility and efficacy of the iEAT manual when it is used in the home home environment with caregivers.

DETAILED DESCRIPTION:
The purpose of the current study is to further develop the integrated Eating Aversion Treatment (iEAT) manual and address the unmet needs of many children with chronic food refusal by providing a technology-based treatment that makes it easy for parents to understand how to duplicate the models of institutional care. The study seeks to expand upon this treatment by introducing the manual and procedures in an electronic form to be implemented by caregivers in a home environment.

The study team aims to enroll 20 participants with chronic food refusal and formula or feeding tube dependence. Participants will be randomly assigned to receive the iEAT manual intervention with the technology supported manual or a control group (10 participants per group). The intervention with the iEAT manual will involve 10 biweekly outpatient appointments of about 45 minutes in length. Target behaviors will be assessed during each treatment meal. Participants will be assessed pre-treatment and at a one month follow-up to assess long term effects. Parents in the control group will provide a food diary once a month, for 5 months. Those assigned to the control group will be able to cross-over to receive the iEAT treatment manual following completion of post-study measures. Screening, collecting data for outcomes measures, and the intervention will be conducted at the each participant's home. Data will be collected on parent compliance with the treatment manual and child food acceptance, nutritional intake, and refusal behaviors.

ELIGIBILITY:
Inclusion Criteria, for the child:

* The child demonstrates failure to meet appropriate nutritional and/or energy needs based on Diagnostic and Statistical Manual (DSM)-V criteria (American Psychiatric Association, 2013) for Avoidant/Restrictive Food Intake Disorder
* Present with partial food refusal as evidenced by greater than 50% of caloric needs met by bottle, formula, or tube feedings
* Have a medical history significant for an organic factor (e.g., gastrointestinal issues) which precipitated or played a role in the development of feeding concern

Inclusion Criteria, for the parent/caretaker:

* Must be English literate
* Must have access to an iPad or a computer

Exclusion Criteria, for the child:

* Patients with active medical diagnoses requiring hospitalization or significant oversight from a physician
* Patients with active medical, structural, or functional limitations preventing safe oral intake of pureed foods (e.g., aspiration, upper airway obstruction)

Exclusion Criteria, for the parent/caretaker:

* Caregivers do not commit to implementing the structured feeding protocol at least 2 times daily

Ages: 12 Months to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Change in acceptance of food during a 10-minute meal | Baseline, end of follow-up (up to 22 weeks)
  A 10-minute meal observation to measure outcomes: acceptance, swallowing, disruption and grams consumed will be rated by trained observers using conventions established in our Feeding Disorders Program. This data collection system will also be used to record child and parent behaviors during outpatient therapy appointments to guide feedback.

SECONDARY OUTCOMES:
Change in disruptions during a 10-minute meal | Baseline, end of follow-up (up to 22 weeks)
  A 10-minute meal observation to measure outcomes: acceptance, swallowing, disruption and grams consumed will be rated by trained observers using conventions established in our Feeding Disorders Program. This data collection system will also be used to record child and parent behaviors during outpatient therapy appointments to guide feedback.
Change in grams of food consumed during a 10-minute meal | Baseline, end of follow-up (up to 22 weeks)
  A 10-minute meal observation to measure outcomes: acceptance, swallowing, disruption and grams consumed will be rated by trained observers using conventions established in our Feeding Disorders Program. This data collection system will also be used to record child and parent behaviors during outpatient therapy appointments to guide feedback.
Change in Clinical Global Impression - Improvement scale (CGI-I) score | Baseline, end of follow-up (up to 22 weeks)
  The Clinical Global Impression - Improvement (CGI-I) scale is a seven-point scale measuring overall change from baseline. Scores will be ranked from 1 (Very Much Improved) through 4 (Unchanged) to 7 (Very Much Worse). Scores of "Much Improved" or "Very Much Improved" will be used to define positive responses; all other scores will indicate negative responses.
Change in Parenting Stress Index-Short Form (PSI) score | Baseline, end of follow-up (up to 22 weeks)
  The Parenting Stress Index-Short Form (PSI) is a 36-item survey commonly used will measure parental stress.

CONTACTS AND LOCATIONS:
Overall Officials: William Sharp, PhD, Principal Investigator — Emory University
Locations (1):
- Marcus Autism Center, Atlanta, Georgia, United States